CLINICAL TRIAL: NCT03435029
Title: Comprehensive Cognitive Remediation as a Strategy to Prevent Cognitive Impairment Associated With Age and Disability in the Elderly With the REHACOP Program
Brief Title: Comprehensive Cognitive Remediation as a Strategy to Prevent Cognitive Impairment Associated With Age and Disability With the REHACOP Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Deusto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: NSMC-004-UD
Record Dates: First submitted 2018-01-26; First posted 2018-02-15 (Actual); Last update posted 2019-07-18 (Actual); Status verified 2019-07

CONDITIONS: Aging
Keywords: aging; cognitive rehabilitation; REHACOP
MeSH Terms: interventions — Occupational Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive Remediation Program (REHACOP) (Experimental): The cognitive rehabilitation program (REHACOP) is a 5 month intervention that allows both individual and group intervention. For the purpose of this study, we included intervention in several domains: attention, language, memory, processing speed, and executive functioning for 3 months, 3 times per week, in 60 minute per session.
  Interventions: Behavioral: Cognitive Remediation Program (REHACOP)
- Occupational Therapy (Active Comparator): The control group performed of occupational group activities (memory tasks, reading the newspaper, drawing, singing or doing crafts). These activities were accomplished in a group format and with the same frequency as the implementation of REHACOP in the experimental group.
  Interventions: Other: Occupational Therapy

INTERVENTIONS:
Behavioral: Cognitive Remediation Program (REHACOP) — The REHACOP group received cognitive remediation sessions 3 times per week for 3 months in 60 minute per session. The rehabilitation consisted of 39 sessions divided into: attention and concentration unit (sustained, selective, alternating, and divided attention) 4 weeks; learning and memory unit (verbal and visual memory and learning strategies) 3 weeks; language (verbal fluency, syntax, grammar, vocabulary, and comprehension) 3 weeks; and executive functioning (objectives planning and attainment, verbal reasoning, categorization, and conceptualization). In addition, processing speed was trained transversely during all the sessions.
  Arms: Cognitive Remediation Program (REHACOP)
Other: Occupational Therapy — The control group received occupational group activities (reading the newspaper, drawing, singing or doing crafts) with the same frequency and format as the experimental group.
  Arms: Occupational Therapy

SUMMARY:
The aim of the study was to analyze the effectiveness of a comprehensive cognitive remediation program (REHACOP) in the non demented elderly, obtaining improvements in cognition and functional skills. It was a longitudinal randomized controlled trial with three assessments: basal, post-treatment, and 12-month follow-up.

Recruitment and enrollment were conducted between September 2012 and November 2016. All participants underwent a clinical interview and an extensive neuropsychological battery. Patients were randomized in an experimental and a control group. The groups were formed by a maximum of eight participants run by an experienced therapist. The experimental group received cognitive remediation for 3 months, 3 times per week, 60 minutes per session. The control group consisted of occupational group activities (reading the newspaper, drawing, singing or doing crafts) with the same frequency as the experimental group. Post-treatment assessment was carried out within the first week after completing the intervention. Finally, longitudinal follow-up at 12 months with neuropsychological assessments will be performed.

Objective: To examine the efficacy of a comprehensive cognitive training program (REHACOP) to improve cognition, clinical symptoms and functional disability for the elderly.

DETAILED DESCRIPTION:
- Neuropsychological assessment

Premorbid IQ was tested by the following tests:

* Accentuation Reading Test (TAP). This test estimates the premorbid IQ in Spanish speakers through 30 words without accentuation which must be read considering its accentuation. Maximum score of 30 points with higher scores indicating better performance.
* Readers assessment processes (PROLEC) (Pseudoword reading). Evaluates the reading ability and the processes that in it intervene. It consists of 40 pseudowords that must be read correctly as quickly as possible. The scores range from 0 to 40. Higher scores indicate better performance.
* Cognitive Reserve Questionnaire (CRQ). This questionnaire consists of fifteen items that measure the cognitive reserve and includes questions about education/culture, working activity, leisure and hobbies, physical activities and social activities. Maximum score of 26 points with higher scores indicating greater cognitive reserve.

Cognitive status was tested by the following tests:

* Mini Mental State Examination (MMSE) determine cognitive status in five categories (orientation, registration, attention and calculation, recall and language). Maximum score of 30 points with higher scores indicating greater performance.
* Montreal Cognitive Assessment (MOCA)* determine cognitive status in nine categories (visuospatial, executive functioning, naming, memory, attention, language, abstraction, delayed recall and orientation). Maximum score of 30 points with higher scores indicating greater performance.

Neurocognitive status was tested by the following tests:

* The Brief Test of Attention (BTA) consists of two parallel forms, numbers and letters, in which the same 10 sequences of random digits and characters were auditory presented at the rate of one stimulus per second. Maximum score of 20 points, 10 points per parallel form. Higher scores indicate greater performance in attention.
* Digit Span Test (WAIS-III). Forward Digits is composed with sixteen series of numbers which have to be repeated in the same order. Maximum score of 16 points with higher scores indicating greater performance. Backward Digits includes fourteen series of numbers have to be repeated backwards. Maximum score of 14 points with higher scores indicating greater performance. These subtests were used to measure attention and working memory.
* Calibrate Ideational Fluency Assessment (CIFA) measures the verbal fluency of words beginning with the letter "p" in three minutes and animals and supermarket categories in 1 minute. Higher number of words indicate better performance.
* Hopkins Verbal Learning Test Revised (HVLT-R) measures performance in verbal memory, learning, and long-term recall in which a list of words is read up to three times (parallel versions 2 and 4 corresponding to basal and post-treatment assessment). Maximum score of 36 points for learning and 12 points for long-term recall with higher scores indicating greater performance.
* Brief Visual Memory Test Revised (BVMT-R) measures performance in visual memory, learning and long-term recall (version 1). Six geometric figures are presented three times. Maximum score of 36 points for learning and 12 points for long-term recall with higher scores indicating greater performance.
* Taylor Complex Figure Test (TCF)* includes 2 conditions (free drawing and copy). The total scores range from 0 to 36 points for each condition with higher scores indicating greater performance in visuoconstructive abilities and visual memory.
* Clock Drawing Test (CDT) is used for screening for cognitive impairment and dementia and as a measure of spatial dysfunction and neglect. This test includes 2 conditions (free drawing and copy). The total scores range from 0 to 10 points for each part with higher scores indicating greater performance.
* Visual Object and Space Perception Battery (VOSP) is a complex battery. Only two subtests have been taken into account, incomplete letters and cube analysis. Higher scores indicating greater performance.
* Trail Making Test (TMT-A, TMT-B). Trail Making Test-A consist of twenty-five numbers have to be ordered from the lowest to the highest in the shortest time possible (i.e., 1-2-3…).Trail Making Test-B consist of alternating between thirteen numbers and twelve letters in an ascending sequence. Shorter time indicates better performance in processing speed and executive functioning.
* Salthouse Perceptual Comparison Test (SPCT) includes two strings of letters that have to be compared and marked as different or equal. Maximum score of 64 points with higher scores indicating greater performance in processing speed.
* Stroop Test is composed of three subtests: word-reading, word-color and interference scores. The examinee has to state the highest number of words or colors in a given time. Higher points indicate greater performance in executive functioning.
* Modified Wisconsin Card Sorting Test (M-WCST)* consists of classifying 48 cards. It is used for evaluating for executive functioning as well as for mental flexibility. The performance of the test will depend on the categories completed correctly, perseverative errors, and total errors.

In order to create a neurocognition composite score, all raw scores were converted to z-scores. The neurocognition composite score was based on the following test and subtest included in the protocol, that is: BTA total score, total score of the forward digits and total score of the backward digit of the WAIS-III, total number of word beginning with the letter "p" in three minutes and total number of words for animals and supermarket categories in one minute of the CIFA, total score of learning and total score of long-term recall of the HVLT-R, total score of learning and total score of long-term recall of the BVMT-R, total score of the free drawing of the CDT, total score of letters and total score of the cube analysis of the VOSP, time of the TMT-A, total score of the SPCT, and total score of the word-color trial of the Stroop Test.

All raw scores were converted to z-scores. TMT-A score was adjusted so that higher scores indicated better cognitive performance. The z-scores were pooled into composite score with the average of the tests and subtest mentioned above.

- MOCA*, TCF*, and M-WCST* tests were added to the protocol after starting the study. TCF and M-WCST were not included to calculate the neurocognition composite score.

Clinical variables, functional variables and subjective complaints were measured by the following tests. Raw scores were used in order to facilitate clinical interpretation.

* Geriatric Depression Scale (GDS-15) includes 15 items. Higher scores indicate a higher degree of depression (range from 0 to 15 points).
* Neuropsychiatric Inventory Questionnaire (NPI-Q) includes 10 neuropsychiatric domains (delusions, hallucinations, agitation/aggression, depression/dysphoria, anxiety, euphoria, apathy, disinhibition, irritability, and aberrant motor behavior) assessed in terms of severity and frequency in a range from 0 to 120 points. Higher scores indicate greater neuropsychiatric behaviors.
* Lille Apathy Rating Scale (LARS) is composed by 33 items, subdivided into 9 subscales (everyday productivity, interests, taking initiative, novelty seeking/motivation, emotional responses, concern, social life, and self-awareness). These subscales are summed into a total score with a possible range from -36 to 36 points. Lower scores indicate a higher degree of apathy.
* Multidimensional Fatigue Inventory (MFI) is composed by 20 items divided into 5 subscales (general index, physical fatigue, mental fatigue, lack of motivation, lack of activity). Higher scores indicate greater fatigue (range from 0 to 140 points).
* Satisfaction With Life Scale (SWLS). This scale is composed by 5 items. Higher scores indicate greater live satisfaction (range from 0 to 35 points).
* Subjective complains were assessed by Subjective Questionnaire on Cognitive and Functional Complains of the patient and caregivers. These questionnaires are composed by 40 items each one of them. Higher scores indicate greater subjective complains (range from 0 to 120 points).

  * Description of the intervention

REHACOP is a comprehensive cognitive remediation program structured in cognitive domains and three levels of difficulty. It is theoretically based on strategies of cognitive rehabilitation (restoration, compensation and optimization). REHACOP uses mainly a bottom-up approach in such a way that it begins with the simplest cognitive domains and ends with the most complex domains and top-down strategies to help with generalization of abilities in daily life. It contains more than 300 paper and pencil tasks, hierarchically structured in 4 modules of cognition (attention and concentration, learning and memory, language and executive functioning), 3 modules of functionality (social cognition, social skills and activities of daily living) and a module of psychoeducation. In this study we used a modified version of REHACOP for the elderly. The REHACOP group received cognitive remediation sessions 3 times per week for 3 months 60 minutes per session. The remediation sessions were performed in the actual homes for the elderly. The groups were made up of a maximum of 8 participants. In particular, the rehabilitation of the REHACOP group consisted of 39 sessions divided into: attention and concentration unit (sustained, selective, alternating, and divided attention) 4 weeks; learning and memory unit (verbal and visual memory and learning strategies) 3 weeks; language (verbal fluency, syntax, grammar, vocabulary, and comprehension) 3 weeks; executive functioning (objectives planning and attainment, verbal reasoning, categorization, and conceptualization) and processing speed were trained transversely during the sessions. This study did not apply the remaining modules (social cognition, social skills, daily living activities and psychoeducation).

ELIGIBILITY:
Inclusion Criteria:

1. age over 55 years
2. signing informed consent
3. independence in daily living activities

Exclusion Criteria:

1. history of neurological or psychiatric conditions, Neuropsychiatric Inventory Cummings > 4
2. illiterate
3. Mini Mental State Examination < 20
4. severe physical constraints.

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2012-09 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Change from baseline to post-treatment and follow-up on one final neurocognition composite score after receiving cognitive remediation. | 3 months and 12 months follow-up
  The neurocognition composite score is one z score that was based on the following test: BTA total score, total score of the forward digits and backward digit of the WAIS-III, total number of words beginning with the letter "p" in 3-minute and total number of words for animals and supermarket categories in 1-minute of the CIFA, total score of learning and total score of long-term recall of the HVLT-R, total score of learning and long-term recall of the BVMT-R, total score of the free drawing of the CDT, total score of letters and total score of the cube analysis of the VOSP, time of the TMT-A, total score of the SPCT, and total score of the word-color trial of the Stroop Test. All raw scores were converted to z-scores. TMT-A score was adjusted so that higher scores indicated better performance. The z-scores were pooled into one composite score with the average of the primary measures mentioned above. Higher scores in this composite score indicated better performance.

SECONDARY OUTCOMES:
Change from baseline score to post-treatment and follow-up on Geriatric Depression Scale (GDS) | 3 months and 12 month follow-up
  Geriatric Depression Scale (GDS-15) includes 15 items. Higher scores indicate a higher degree of depression (range from 0 to 15 points).
Change from baseline score to post-treatment and follow-up on Neuropsychiatric Inventory Questionnaire (NPI-Q) | 3 months and 12 months follow-up
  Neuropsychiatric Inventory Questionnaire (NPI-Q) includes 10 neuropsychiatric (delusions, hallucinations, agitation/aggression, depression/dysphoria, anxiety, euphoria, apathy, disinhibition, irritability, and aberrant motor behavior) domains assessed in terms of severity and frequency in a range from 0 to 120 points. Higher scores indicate greater neuropsychiatric behaviors.
Change from baseline score to post-treatment and follow-up on Lille Apathy Rating Scale (LARS) | 3 months and 12 months follow-up
  Lille Apathy Rating Scale (LARS) is composed by 33 items, subdivided into 9 subscales (everyday productivity, interests, taking initiative, novelty seeking/motivation, emotional responses, concern, social life, and self-awareness). These subscales are summed into a total score with a possible range from -36 to 36 points. Lower scores indicate a higher degree of apathy.
Change from baseline score to post-treatment and follow-up on Multidimensional Fatigue Inventory (MFI) | 3 months and 12 months follow-up
  Multidimensional Fatigue Inventory (MFI) is composed by 20 items divided into 5 subscales (general index, physical fatigue, mental fatigue, lack of motivation, lack of activity). Higher scores indicate greater fatigue (range from 0 to 140 points).
Change from baseline score to post-treatment and follow-up on Satisfaction With Life Scale (SWLS) | 3 months and 12 months follow-up
  Satisfaction With Life Scale (SWLS). This scale is composed by 5 items. Higher scores indicate greater live satisfaction (range from 0 to 35 points)
Change from baseline score to post-treatment and follow-up on Subjective Questionnaire on Cognitive and Functional Difficulties of the patient and caregivers | 3 months and 12 months follow-up
  Subjective complains were assessed by Subjective Questionnaire on Cognitive and Functional Complains of the patient and caregivers. These questionnaires are composed by 40 items each one of them. Higher scores indicate greater subjective complains (range from 0 to 120 points).

CONTACTS AND LOCATIONS:
Overall Officials: Natalia Ojeda del Pozo, PhD, Principal Investigator — University of Deusto
Locations (1):
- University of Deusto, Bilbao, Bizcay, Spain

REFERENCES:
- [Derived] Montoya-Murillo G, Ibarretxe-Bilbao N, Pena J, Ojeda N. Effects of Cognitive Rehabilitation on Cognition, Apathy, Quality of Life, and Subjective Complaints in the Elderly: A Randomized Controlled Trial. Am J Geriatr Psychiatry. 2020 May;28(5):518-529. doi: 10.1016/j.jagp.2019.10.011. Epub 2019 Oct 21. PMID 31735487